CLINICAL TRIAL: NCT05850988
Title: Effects of Different Oxygen Concentrations for Preoxygenation on Lung Ultrasound Scores During Spontaneous Ventilation
Brief Title: Effects of Different Oxygen Concentrations on Lung Ultrasound Score During Spontaneous Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, derya özkan, Professor M.D., Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: AESH-EK1-2023-001
Record Dates: First submitted 2023-04-06; First posted 2023-05-09 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Atelectasis
Keywords: atelectasis; preoxygenation; lung ultrasound; general anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Eighty (Active Comparator): Patients in Group E will receive %80 oxygen for 3 minutes during preoxygenation
  Interventions: Other: %80 Oxygen concentration
- Group Hundred (Active Comparator): Patients in Group H will receive %100 oxygen for 3 minutes during preoxygenation
  Interventions: Other: %100 Oxygen concentration

INTERVENTIONS:
Other: %80 Oxygen concentration — Patients will be administered %80 Oxygen for 3 minutes during preoxygenation.
  Other Names: %80 Inspired fraction of oxygen
  Arms: Group Eighty
Other: %100 Oxygen concentration — Patients will be administered %100 Oxygen for 3 minutes during preoxygenation.
  Other Names: %100 Inspired fraction of oxygen
  Arms: Group Hundred

SUMMARY:
The goal of this study is to observe the effects of different oxygen concentrations during preoxygenation in spontaneous breathing patients with modified lung ultrasound scores before induction of general anesthesia. Preoxygenation is a routine and recommended procedure for patients undergoing general anesthesia. Atelectasis is a common side effect of general anesthesia and usage of high concentration oxygen is a probable cause of it. Using lower oxygen concentrations in preoxygenation may help reducing the atelectasis and it can be assessed by lung ultrasound.

DETAILED DESCRIPTION:
Preoxygenation is the process of supplying the patient a high inspired fraction of oxygen prior to an airway intervention or induction of general anesthesia. Prolonging safe apnea duration is the primary aim of preoxygenation and preoxygenation is recommended for all patients before induction of general anesthesia.

Atelectasis is the most common postoperative pulmonary complication and is associated with usage of high inspired fraction of oxygen. Modified lung ultrasound scoring is an effective and noninvasive method to determine atelectasis. In this study we will observe the effects of different oxygen concentrations during preoxygenation before induction of general anesthesia in spontaneous breathing patients with modified lung ultrasound scores .

Patients undergoing general anesthesia for elective surgery meeting the criteria will be acknowledged about the study. After written consents are taken patients will be randomised into two groups by coin method. One group will receive %80 oxygen for 3 minutes and other group will receive %100 oxygen for 3 minutes during preoxygenation. Each participants demographic data will be collected. 12 quadrants of thorax divided by midsternal line, anterior axillary and posterior axillary lines will be examined by the usage of modified lung ultrasound score before and at the end of preoxygenation for all individuals. Randomisation, lung ultrasound scoring and preoxygenation will be done by different experienced anesthesiologists so the observers of this study would be blinded for the results. Patients will be blinded for the concentration of oxygen. Modified lung scores of each group would be compared at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Score I and II
* Being a candidate to elective surgery under general anesthesia

Exclusion Criteria:

* Patients with any pulmonary disease
* Patients who had pulmonary infection in the past 3 months
* Patients who had a surgery in the past 3 months
* Patients who had a multitrauma in the past 3 months
* Patients who have a Body Mass Index over 30
* Pregnants
* Patients who have diaphragma hernia
* Patients who have gastroesophageal reflux disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change of Modified Lung Ultrasound Scores | 3 minutes
  Scores between 0-3 for 12 thorax quadrants and total score will be recorded for each participants before and after a 3 minutes time of preoxygenation to assess change from baseline

SECONDARY OUTCOMES:
End-Tidal Oxygen levels | 3 minutes
  End-tidal oxygen levels at the end of 3 minutes of preoxygenation will be recorded for each participants

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozkan, Professor MD, Principal Investigator — Ozkan D
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555